CLINICAL TRIAL: NCT02054507
Title: Prematurity Related Risks of Cognitive Impairment at School Age With Regards to Social, Family and Care Environment
Brief Title: Prematurity Related Risks of Cognitive Impairment at School Age
Acronym: NEORIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean Michel Hascoet (Other)
Collaborators: Maternite Regionale Universitaire (Other)
Responsible Party: Sponsor-Investigator, Jean Michel Hascoet, Professor, Maternite Regionale Universitaire
Organization: Maternite Regionale Universitaire (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRU.10.11; NEORIS (Other: Maternite Regionale Universitaire)
Record Dates: First submitted 2014-01-27; First posted 2014-02-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Complications of Prematurity
Keywords: Children; Cognitive outcome; Prematurity; Care Network; Outpatient follow-up of cognitive development; Care resources
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Former premature infants (No Intervention): Cognitive and executive evaluation by Wechsler IV tests
  Interventions: Behavioral: Cognitive evaluation (Wechsler IV tests)

INTERVENTIONS:
Behavioral: Cognitive evaluation (Wechsler IV tests) — Children born prematurely in a level III referral Center will undergo psychometric evaluation at 8 to 11 years of age by routine test (WISC IV). The relationship between cognitive scores and neonatal characteristics will be determined and compared with the results of schoolmate control children, born at term.

SUMMARY:
The main purpose of this study is to better evaluate prematurely born children cognitive development at school age, with regards to birth conditions but also to social situation, intra family relationships, and modalities of care.

The study will be divided into 3 parts:

1. Children born prematurely in our level III referral Center will undergo psychometric evaluation at 8 to 11 years of age by routine cognitive test. The relationships between cognitive scores and neonatal characteristics will be determined and compared to the results of schoolmates born at term.
2. The quality of parent and child relationship will be evaluated by a standardized questionnaire allowing the evaluation of persistent stress trauma related to premature birth.
3. An anthropologic study of the utilization of care resources will also be performed within the follow-up network taking care of these children.

DETAILED DESCRIPTION:
Long term follow-up of vulnerable children such as infants born prematurely are generally studied without taking into account the social, familial and care resources available in the child environment.

Thus, the main purpose of this study is to evaluate prematurely born children cognitive development at school age, with regards to birth conditions but also to related social situation, intra family relationships, modalities of care and utilization of care resources.

The study will be divided into 3 parts:

1. Children born prematurely in our level III referral Center will undergo psychometric evaluation at 8 to 11 years of age by routine test (WISC IV). The relationship between cognitive scores and neonatal characteristics will be determined and compared with the results of schoolmate control children, born at term.
2. The quality of parent and child relationship will be evaluated by standardized questionnaire (Perinatal PTSD Questionnaire). This questionnaire allows evaluating persistent perinatal stress trauma related to prematurity.
3. An anthropologic study of care and utilization of care resources will be performed within the follow-up network taking care of these children. This part will use semi-directive interviews of caregivers involved in the follow-up network.

This study should allow to better correlate prematurely born children outcome with their global environment and propose improvements in care resources utilization for a better development.

ELIGIBILITY:
Inclusion Criteria:

* Former premature infants aged 8-11 years
* School grade appropriate for their age
* Schoolmate control children born at term aged 8-11 years

Exclusion Criteria:

* Any neurological sequelae

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cognitive and executive functions at school age in prematurely born children | Children at the age of 8-11 years
  Assessment by WECHSLER IV tests of children born prematurely without neurological or sensorial sequelae, and without psychological difficulties; All in school grade appropriate for their ages
  Controls : children born at term, matched for age and school grade.

SECONDARY OUTCOMES:
Quality of parent and children relationship | Evaluated at 8-11 years of children (at the time of child cognitive evaluation)
  Evaluation will be performed by standardized questionnaire (Perinatal PTSD Questionnaire). This questionnaire allows evaluating persistent perinatal stress trauma related to prematurity.

OTHER OUTCOMES:
Utilization of care resources | Evaluation of care network up to 18 months (within the time for children cognitive evaluation)
  anthropologic study of care and utilization of care resources using semi-directive interviews of caregivers involved in the follow-up network

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, Principal Investigator — Maternite Regionale Universitaire CHU NANCY
Locations (2):
- France (2):
  - M.S.H. Lorraine/Lorraine Institue for Social Sciences and Humanities (CNRS, Université de Lorraine), Nancy
  - Maternite Regionale Univesitaire, Nancy